CLINICAL TRIAL: NCT00890305
Title: Phase II Study to Evaluate the Safety, Tolerability and Efficacy of FOLFOX + CT-011 Versus FOLFOX Alone Administered Intravenously to Patients With Colorectal Adenocarcinoma Previously Untreated for Metastatic Disease
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of FOLFOX + CT-011 Versus FOLFOX Alone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-2008-01; 2009-014593-18 (EudraCT Number)
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; FOLFOX chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pidilizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-011 in combination with FOLFOX (Experimental): CT-011 (3 mg/kg) administered intravenously every 4 weeks for 4 weeks and every 12 weeks thereafter until disease progression or maximum tolerance.
  FOLFOX (FOLFOX4 or mFOLFOX6) administered 7 days after the first administration of CT-011 and repeated every 14 days for up to 24 cycles. At the end of FOLFOX therapy, patients who have not progressed will be eligible for maintenance chemotherapy with 5-FU/leucovorin at the same dose and schedule until disease progression or study drug discontinuation.
  Interventions: Drug: CT-011; Drug: FOLFOX
- FOLFOX (Active Comparator): FOLFOX (FOLFOX-4 or mFOLFOX6) administered every 14 days for up to 24 cycles. At the end of FOLFOX therapy, patients who have not progressed will be eligible for maintenance chemotherapy with 5-FU/leucovorin at the same dose and schedule until disease progression or study drug discontinuation.
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: CT-011
  Arms: CT-011 in combination with FOLFOX
Drug: FOLFOX — FOLFOX-4: each cycle consists of the following: oxaliplatin 85 mg/m2 on Day 1, leucovorin 200 mg/m2/day on Day 1 and Day 2 followed by 5-FU 400 mg/m2 bolus and a 22 hour infusion of 5-FU 600 mg/m2 for two consecutive days.
  mFOLFOX-6: each cycle consists of the following: oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 on Day 1, followed by 5-FU 400 mg/m2 bolus, followed by 5-FU 1200 mg/m2/day for two consecutive days (total 2,400 mg/m2 over 46-48 hours).

SUMMARY:
This clinical trial will be performed in previously untreated patients with metastatic colorectal cancer. The study will evaluate the safety, tolerability and efficacy of the study drug, CT-011, in combination with FOLFOX chemotherapy (FOLFOX4 or mFOLFOX6) compared with treatment by FOLFOX alone.

DETAILED DESCRIPTION:
The proposed clinical trial will be a multi-center, randomized, open label, active control study in previously untreated patients with metastatic colorectal cancer aimed to evaluate the safety, tolerability and efficacy of the monoclonal antibody, CT-011, administered at 3mg/kg in combination with FOLFOX chemotherapy (FOLFOX4 or mFOLFOX6) compared with treatment by FOLFOX alone. Approximately 168 patients are planned to be enrolled to this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is 18 years or older, both genders.
2. Patients with metastatic disease who are eligible for first line FOLFOX chemotherapy. Adjuvant or neoadjuvant given at least 12 months prior for non-metastatic disease is permitted.
3. ECOG performance status ≤ 1
4. At least 4 weeks from prior major surgery or radiotherapy.
5. Life expectancy >3 months
6. Hematology: ANC ≥ 1.5X109/L; Platelets >100x109/L.
7. Adequate Renal function
8. Adequate Hepatic functions
9. Normal Cardiac function

Exclusion Criteria:

1. Patients who had adjuvant or neoadjuvant therapy for non-metastatic disease given within the last 12 months.
2. Patients who had received Oxaliplatin within 12 months prior to diagnosis of metastatic disease.
3. Patients on concurrent anti cancer therapy other than that allowed in the study.
4. Patients on concurrent steroids, other than those allowed for routine antiemetics, or inhaled steroids
5. Presence of clinically apparent or suspected brain metastasis.
6. Patients who have had myocardial infarction, severe congestive heart failure, or significant arrhythmia within the past 6 months.
7. Serious active infection at the time of pre-study screening.
8. Active or history of autoimmune disorders/conditions.
9. Women who are pregnant or lactating
10. Concurrent active malignancy.
11. Ascites, pleural effusions, or osteoblastic bone metastases as the only site of disease.
12. Other prior malignancies, except for cured or adequately treated malignancies for which there has been no evidence of activity for more than 5 years.
13. Subjects with a condition which may interfere with the subjects' ability to understand the requirements of the study.
14. Patients with history of life threatening allergic reactions to food or drugs
15. Patients with symptomatic peripheral neuropathy> Grade 1.
16. Known positive HIV, Hepatitis B surface antigen or Hepatitis C antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the median progression free survival in patients treated with CT-011 plus FOLFOX compared to that of patients treated with FOLFOX alone. | 32 months

SECONDARY OUTCOMES:
Composite of safety, tolerability, pharmacokinetics and immunogenicity of CT-011. | 32 months
Anti tumor activity of the antibody. | 32 months
Objective response rate by RECIST. | 32 months
Progression-free survival rates. | 32 months
Response duration. | 32 months
Overall survival. | 32 months
Tumor and immunological markers. | 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (31):
- United States (5):
  - The Cancer Center of Huntsville, PC, Huntsville, Alabama
  - University of South Florida, Tampa, Florida
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
- Bulgaria (7):
  - MHAT "Dr. Tota Venkova", Gabrovo
  - InterDistrict Dispensary in Oncology Diseases with Stationary-Ruse, EOOD, Rousse
  - InterDistrict Dispensary in Oncology Diseases with Stationary, Shumen
  - Multiprofile Hospital for Active Treatment "Tsaritza Joanna", Sofia
  - Specialized Hospital for Active Treatment for Oncology, Sofia
  - InterDistrict Dispensary of Oncology Diseases with Stationary, Varna
  - Multiprofile Hospital for Active Treatment "Sv. Marina", EAD,, Varna
- India (6):
  - Regional Cancer Centre, Indira Gandhi Institute of Medical Sciences, Sheikhpura, Patna, Bihar
  - Cancer Clinic, Nagpur, Maharashtra
  - Curie Manavata Cancer Centre, Opp., Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - G. Kuppuswamy Naidu Memorial Hospital, Pappanaickenpalayam, Coimbatore, Tamil Nadu
- Peru (3):
  - Hospital Almanzor Aguinaga Asenjo - Chiclayo, Chiclayo
  - Clinica Ricardo Palma, Lima
  - Hospital Regional nivel III Cayetano Heredia Essalud Piura, Piura
- Puerto Rico (2):
  - Ponce School of Medicine/CAIMED Center, Ponce
  - Fundacion de Investigacion de Diego, Santurce
- Romania (8):
  - "Prof. Dr. Ion Chiricuţă" Institute of Oncology, Cluj-Napoca
  - Clinical Emergency Hospital - Oncology Department, Constanța
  - Oncolab SRL, No. 1, Craiova
  - Center of Medical Oncology, Iași
  - Clinical Hospital Pelican Oradea, Oradea
  - No. 1 City Hospital, Ploieşti
  - "Sf. Ioan cel Nou" Clinical Emergency County Hospital, Suceava
  - Clinic of Oncology - Radiotherapy, Tg. Mures